CLINICAL TRIAL: NCT05738382
Title: A Randomized, Double-blind, Open for Active Comparator, Parallel, Multi-center Phase II Study to Explore the Efficacy, Safety and Tolerability of BG2109 Compared With Cetrorelix During COH in Female Subjects Undergoing ART Procedures
Brief Title: Efficacy and Safety of BG2109 During Controlled Ovarian Hyperstimulation in Female Subjects Undergoing ART Procedures
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bio Genuine (Shanghai) Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BG2109-AC-201
Record Dates: First submitted 2023-01-28; First posted 2023-02-22 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Assisted Reproductive Technology; Controlled Ovarian Hyperstimulation
MeSH Terms: interventions — cetrorelix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masked for BG2109 dose groups and open for the active controlled group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BG2109 75mg (Experimental): oral, once a day
  Interventions: Drug: BG2109
- BG2109 150mg (Experimental): oral, once a day
  Interventions: Drug: BG2109
- BG2109 200mg (Experimental): oral, once a day
  Interventions: Drug: BG2109
- Cetrorelix (Active Comparator): 0.25mg, Subcutaneous injection, once a day
  Interventions: Drug: Cetrorelix

INTERVENTIONS:
Drug: BG2109 — oral administration once daily
  Arms: BG2109 150mg; BG2109 200mg; BG2109 75mg
Drug: Cetrorelix — 0.25 mg, Subcutaneous injection once daily.
  Other Names: Cetrorelix Acetate
  Arms: Cetrorelix

SUMMARY:
To explore the optimal effective daily dose of BG2109 to suppress premature luteinizing hormone (LH) surge during COH in female subjects undergoing ART procedures.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, open for active comparator, parallel, multi-center phase II dose-finding clinical study to explore the efficacy, safety and tolerability of different doses of BG2109 compared with Cetrorelix during Controlled Ovarian Hyperstimulation (COH) in Chinese female subjects undergoing Assisted Reproductive Technology (ART) procedures.

ELIGIBILITY:
Inclusion Criteria:

* Married infertile women aged 20 to 39 years (both inclusive), who are diagnosed with tubal infertility, unexplained infertility, grade I-II endometriosis, or spouses diagnosed with male factor infertility, who meet the criteria for IVF and/or ICSI) using fresh or frozen semen from the male spouse or sperm donor
* BMI 18-25 kg/m2 (both inclusive), body weight range 45-80kg (both inclusive)
* Subjects must have regular menstrual cycles, specifically defined as ≥25 days, ≤35 days.
* The serum sex hormone levels during the screening period must be performed in the early follicular phase, and the basal serum follicle-stimulating hormone (FSH) <10 IU/L, LH, estradiol(E2), prolactin(PRL),testosterone(T) levels are within the laboratory normal range, or the investigator considers them as abnormal but not clinically significant
* The subject is clinically assessed and agree to undergo fresh cycle embryo transfer in the first IVF-ET/ ICSI-Embryo Transfer(ET) cycle, with a maximum of two embryos transferred.
* Within 1 year before randomization, the presence of bilateral ovaries is clearly visible on transvaginal ultrasonography with no significant abnormalities, and appendages are normal. Both ovaries must be available for oocyte retrieval
* Subjects must sign the Informed Consent Form (ICF) and be willing and able to abide by the protocol-specified study procedures

Exclusion Criteria:

* Those who have undergone 2 or more COH of IVF/ICSI-ET before screening, but have not achieved clinical pregnancy.
* Those with previous IVF or ART failure due to sperm/fertilization problems whose related medical condition has not been improved.
* Either subjects or their spouses or both of them are known to carry abnormal chromosomal structures, or patients known to have single-gene genetic diseases or serious diseases with genetic susceptibility requiring Preimplantation Genetic Diagnosis(PGD) before embryo transfer.
* Those with high risk of ovarian hyperstimulation syndrome(OHSS)
* Those with low ovarian function at screening, with at least one of the following: poor ovarian response in the past; less than 6 antral follicles (AFC) with a diameter of < 10 mm seen on bilateral ovary transvaginal ultrasonography at Day2-3 of menstrual cycle; anti-mullerian hormone(AMH) < 1.1 ng/ml.
* Subjects who used gonadotropins for ovarian stimulation or drugs that affect ovarian function within 30 days prior to screening.
* Subjects with abnormal thinprep cytology test(TCT) results that are judged by the investigator as clinically significant and require treatment within 6 months before screening.
* As judged by the investigator, subjects with clinically significant gynecological diseases at screening
* Those previously or prior randomization suffering from the cancer of uterine, ovarian, breast or hypothalamus or pituitary gland.
* Those with a positive serum β-hCG test result at the screening visit or the visit on Day 1 of ovarian stimulation.
* During COH, LH ≥10 U/L, and the LH level was 2.5 times higher than the baseline value before D0 (inclusive).

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Suppression rate of premature LH surge from the treatment of investigational medicinal products(IMP) until the day of human chorionic gonadotropin(hCG) injection | Through the whole period of administration of IMP，about 5-10 days
  LH ≥ 10 IU/L

SECONDARY OUTCOMES:
Ongoing pregnancy rate | At 10 weeks post-embryo transfer
  ongoing pregnancy is defined as at least embryo with heartbeat at 10 weeks post-embryo transfer
The number of oocytes obtained on the day of oocyte retrieval | During the surgery of the oocyte retrieval
Clinical pregnancy rate | On 30-37 days after embryo transfer
  clinical pregnancy is defined as the presence of at least one gestational sac in or outside the uterus during 30-37 days after embryo transfer
Adverse drug events | Through study completion, around 45 weeks.
Pharmacokinetics(PK) endpoints | On the morning of the Second and Third day of BG2109 administration, and the day of hCG injection(about 5-10days after BG2109 administration)
  Plasma concentration of BG2109
Pharmacodynamics(PD) endpoints | 30 minutes before the administration of BG2109 every morning through the whole period of IMP administration，about 5-10 days
  estradiol(E2), luteinizing hormone (LH) and progesterone (P) concentrations at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Liang, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (10):
- China (10):
  - Site No5, Changsha
  - Site No7, Guangzhou
  - Site No9, Haikou
  - Site No4, Hangzhou
  - Site No8, Hohhot
  - Site No6, Linyi
  - Site No10, Shenyang
  - Site No11, Tianjin
  - Site No3, Wuhan
  - Site No2, Zhengzhou

IPD SHARING:
Plan to Share IPD: No